CLINICAL TRIAL: NCT02917980
Title: Multicenter Registry Study of Surgery and Transcatheter Intervention for Structural Heart Diseases
Brief Title: Surgery and Transcatheter Intervention for Structural Heart Diseases
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other); Beijing Anzhen Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: XJ-20160829
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2016-09

CONDITIONS: Data Collecting and Analyzing of Different Treatment of Structural Heart Diseases
Keywords: structural Heart Diseases; surgical treatment; interventional treatment; hybrid treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- surgical treatment: patients with structural heart disease received surgical treatment
- interventional treatment: patients with structural heart disease received interventional treatment
- surgical combined with interventional treatment: patients with structural heart disease received surgical combined with interventional treatment

SUMMARY:
This project aimed to optimize the therapeutic strategy for structural heart disease by choosing optimal treatment, such as,surgical treatment,interventional and surgery combined with interventional hybrid treatment. Thereby improve successful rate of clinical treatment, and establish the guideline for treatment of structural heart disease.At the same time,online registration database for structural heart disease will be established to further data analysis and objective assessment of clinical curative effect for structural heart disease in China.

DETAILED DESCRIPTION:
This project is a 5 years prospective,observational,longitudinal registration study on clinical surgical and interventional treatment of structural heart disease.Firstly,patients with structural heart disease, whom received surgical,interventional or surgery combined with interventional hybrid treatment during Jan. 2015 to Jan. 2020 ,were registrated dynamiclly. And further management and 1 year clinical follow-up,which contains demographic characteristics, clinical manifestations, treatment strategies and prognosis of outcome, were performed on the recruited data.Secondly, this is also a prospective observational study, featured by collecting data through annual follow-up,with the timing at the point of off the hospital,and 1,2,6,9,12 month after hospital discharge,respectively.

The inclusion criteria:

1. atrial septal defect
2. ventricular septal defect
3. patent ductus arteriosis
4. pulmonary stenosis
5. residual leakage after surgical treatment for congenital heart disease
6. coronary artery fistula
7. pulmonary arteriovenous malformations
8. tetralogy of Fallot, and other cyanotic heart disease
9. mitral stenosis and insufficiency
10. tricuspid stenosis and insufficiency
11. aortic stenosis and insufficiency
12. pulmonary stenosis and insufficiency
13. coarctation of aorta
14. paravalvular leakage
15. hypertrophic obstructive heart disease
16. dilated cardiomyopathy
17. structural heart disease need surgery combined with interventional hybrid treatment
18. structural heart disease need surgeryor interventional treatment

The exclusion criteria:

1. primary arrhythmia cardiac disease,like tachycardia and ventricular fibrillation
2. circulation disease, like coronary heart disease,hypertension,arterial aneurysm
3. patients were not received any treatment
4. patients were hard to follow-up
5. no informed Consent

ELIGIBILITY:
Inclusion Criteria:

1.atrial septal defect 20ventricular septal defect 3.patent ductus arteriosis 4.pulmonary stenosis 5.residual leakage after surgical treatment for congenital heart disease 6.coronary artery fistula 7.pulmonary arteriovenous malformations 8.tetralogy of Fallot, and other cyanotic heart disease 9.mitral stenosis and insufficiency 10.tricuspid stenosis and insufficiency 11.aortic stenosis and insufficiency 12.pulmonary stenosis and insufficiency 13.coarctation of aorta 14.paravalvular leakage 15.hypertrophic obstructive heart disease 16.dilated cardiomyopathy 17.structural heart disease need surgery combined with interventional hybrid treatment 18.structural heart disease need surgeryor interventional treatment

Exclusion Criteria:

1. primary arrhythmia cardiac disease,like tachycardia and ventricular fibrillation
2. circulation disease, like coronary heart disease,hypertension,arterial aneurysm
3. patients were not received any treatment
4. patients were hard to follow-up
5. no informed Consent

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with structural heart disease, whom received surgical,interventional or surgery combined with interventional hybrid treatment
Sampling Method: Non-Probability Sample
Enrollment: 883 (Actual)
Dates: Start 2016-01; Primary Completion 2020-01 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Death from any cause | 12 months
Cumulative MACE | 12 months
  Cumulative MACE (including death, rupture, paraplegia, aneurysm formation et al)

SECONDARY OUTCOMES:
Acute or chronic renal insufficiency | 12 months
residual shunt or regurgitation | 12 months
cerebral incidence | 12 months
hemolysis | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaan'xi Province, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mao Y, Liu Y, Zhai M, Jin P, Chen F, Yang Y, Zhang G, Shang X, Jian Z, Zhang H, Wei L, Liu J, Guo Y, Pan X, Wu Y, Piazza N, Yang J. Treatment options for young patients with asymptomatic severe aortic stenosis: a multicenter retrospective cohort study. Eur J Med Res. 2025 Oct 14;30(1):966. doi: 10.1186/s40001-025-03227-6. PMID 41088494
- [Derived] Liu Y, Xu C, Jin P, Zhai M, Tang H, Tian Z, Wen A, Qiao R, Yang J. Transcatheter closure of paravalvular leakage through multiple approaches after surgical mechanical valve replacements: A retrospective study. Medicine (Baltimore). 2024 Nov 22;103(47):e40600. doi: 10.1097/MD.0000000000040600. PMID 39809196
- [Derived] Wang Y, Ma Y, Liu Y, Yang J. First Experience With a Novel Self-Expandable Valve for Mitral Annular Calcification Guided by Three-Dimensional Printing. Catheter Cardiovasc Interv. 2025 Mar;105(4):855-860. doi: 10.1002/ccd.31405. Epub 2025 Jan 7. PMID 39763352
- [Derived] Jin P, Guo H, Mao Y, Zhai M, Liu Y, Yang J. Transcatheter mitral valve replacement to treat rheumatic mitral stenosis: a case series. Front Cardiovasc Med. 2024 Dec 5;11:1424105. doi: 10.3389/fcvm.2024.1424105. eCollection 2024. PMID 39703883
- [Derived] Mao Y, Liu Y, Zhai M, Jin P, Zhang H, Wei L, Shang X, Guo Y, Pan X, Yang J. Prognostic value of right ventricular dysfunction in aortic regurgitation after transcatheter aortic valve replacement. Front Cardiovasc Med. 2024 Aug 30;11:1424116. doi: 10.3389/fcvm.2024.1424116. eCollection 2024. PMID 39280033
- [Derived] Li L, Wang Y, Jin P, Yang T, Zhu G, Li Y, Tang J, Liu Y, Yang J. Hemodynamics in the treatment of pseudoaneurysm caused by extreme constriction of aortic arch with coated stent. Front Cardiovasc Med. 2024 Aug 20;11:1363230. doi: 10.3389/fcvm.2024.1363230. eCollection 2024. PMID 39228660
- [Derived] Mao Y, Ma Y, Zhai M, Li L, Jin P, Liu Y, Yang J. Preliminary Study of a Degenerated Tricuspid Bioprosthetic Valve Implanted via Transcatheter Valve-in-Valve Implantation Guided by 3-Dimensional Printing. CJC Open. 2023 Dec 5;6(8):978-988. doi: 10.1016/j.cjco.2023.11.023. eCollection 2024 Aug. PMID 39211748
- [Derived] Wang Y, Liu Y, Meng X, Zhai M, Jin P, Lu F, Yang J. Comparing outcomes of transcatheter tricuspid valve replacement and medical therapy for symptomatic severe tricuspid regurgitation: a retrospective study. Eur J Med Res. 2024 Aug 5;29(1):407. doi: 10.1186/s40001-024-01947-9. PMID 39103966
- [Derived] Mao Y, Liu Y, Zhai M, Yang J. Application of and Prospects for 3-Dimensional Printing in Transcatheter Mitral Valve Interventions. Rev Cardiovasc Med. 2023 Feb 14;24(2):61. doi: 10.31083/j.rcm2402061. eCollection 2023 Feb. PMID 39077424
- [Derived] Chen H, Mao Y, Xie H, Liu D, Zhang S, Tian Y, Yang J, Bai B. Case report: Cardiac metastatic uterine intravenous leiomyomatosis excision with extracorporeal venous shunt under the guidance of 3-dimensional printing. Front Cardiovasc Med. 2023 Jun 15;10:1117227. doi: 10.3389/fcvm.2023.1117227. eCollection 2023. PMID 37396586
- [Derived] Mao Y, Liu Y, Meng X, Ma Y, Li L, Zhai M, Jin P, Lu F, Yang J. Treatment of severe tricuspid regurgitation induced by permanent pacemaker lead: Transcatheter tricuspid valve replacement with the guidance of 3-dimensional printing. Front Cardiovasc Med. 2023 Mar 22;10:1030997. doi: 10.3389/fcvm.2023.1030997. eCollection 2023. PMID 37034329
- [Derived] Liu Y, Zhai M, Mao Y, Xu C, Ma Y, Li L, Jin P, Yang J. Transcatheter aortic valve replacement in patients with quadricuspid aortic valve in a single center. Front Cardiovasc Med. 2022 Sep 28;9:1011466. doi: 10.3389/fcvm.2022.1011466. eCollection 2022. PMID 36247444
- [Derived] Mao Y, Liu Y, Ma Y, Jin P, Li L, Yang J. Mitral Valve-in-Valve Implant of a Balloon-Expandable Valve Guided by 3-Dimensional Printing. Front Cardiovasc Med. 2022 May 30;9:894160. doi: 10.3389/fcvm.2022.894160. eCollection 2022. PMID 35711355
- [Derived] Xu C, Liu Y, Zhai M, Jin P, Li L, Ma Y, Yang J. Transcatheter Closure of a Paravalvular Leak Guided by Transesophageal Echocardiography and Three-Dimensional Printing. Front Cardiovasc Med. 2022 May 20;9:750896. doi: 10.3389/fcvm.2022.750896. eCollection 2022. PMID 35669478
- [Derived] Ding P, Xu C, Liu Y, Meng X, Jin P, Tang J, Li L, Ma Y, Yang J. Application of three-dimensional transesophageal echocardiography in preoperative evaluation of transcatheter aortic valve replacement. BMC Cardiovasc Disord. 2021 Jun 28;21(1):315. doi: 10.1186/s12872-021-02101-7. PMID 34182931
- [Derived] Liu Y, Xu C, Ding P, Tang J, Jin P, Li L, Chen M, Meng X, Zhao H, Yang J. Transcatheter Closure of Mitral Paravalvular Leak via Multiple Approaches. J Interv Cardiol. 2021 Mar 2;2021:6630774. doi: 10.1155/2021/6630774. eCollection 2021. PMID 33746639